CLINICAL TRIAL: NCT00870220
Title: Initiating Transdermal Estradiol Therapy in Turner's Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Collaborators: Novo Nordisk A/S (Industry); University of Michigan (Other); Johns Hopkins University (Other); Massachusetts General Hospital (Other); University of Oklahoma (Other); University of South Florida (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 15327B
Record Dates: First submitted 2009-03-05; First posted 2009-03-27 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Turner's Syndrome
Keywords: Turner's Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone; Estradiol; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GH alone, Low dose E2 patch, Very Low-dose E2 patch (Experimental): Group 1: Growth hormone alone, no E2. Group 2: Growth Hormone plus Estradiol patch dose A(14 mcg/d x 10 d) x 6 months then Estradiol patch dose B(25 mcg/d x 10 d) x 6 months.
  Group 3: Growth Hormone plus Estradiol patch dose B(25 mcg/d x 10 d) x 6 months then Estradiol patch dose C(25 mcg/d x 3 w) x 6 months.
  Interventions: Drug: Norditropin, Menostar 14mcg patch, Vivelle dot 25mcg patch

INTERVENTIONS:
Drug: Norditropin, Menostar 14mcg patch, Vivelle dot 25mcg patch — GH will be maintained at 0.05mg/kg/d, adjusted every 3 months. Estradiol 14mcg patch will be applied for 10 days/month for the first 6 months in Group 2. Estradiol 25mcg patch will be applied for 10 days/month for the second 6 months in Group 2, and for the first 6 months in Group 3. Estradiol 25mcg patch will be applied for 3 weeks per month for the second 6 months in Group 3.
  Other Names: Norditropin; Menostar patch; Vivelle dot patch

SUMMARY:
This is a multicenter, randomized, controlled, semi-blinded study to compare two low doses of estradiol administered by recently available transdermal patches for the initiation of puberty in Turner syndrome girls 11.5-13.0 years old in conjunction with growth hormone (GH) therapy.

The specific hypotheses to be tested are: when combined with growth hormone (GH) treatment, low dose transdermal estradiol (LTE2) replacement will be more effective in stimulating feminization, height velocity, and bone mineral density without compromising growth potential than very low dose transdermal estradiol (VLTE2), which will in turn be superior to GH alone in effects on feminization, height velocity, and bone mineral density.

DETAILED DESCRIPTION:
Determining the estrogen replacement regimen which is optimal with GH therapy is an important issue in the management of Turner syndrome today. The estrogen effect on growth is biphasic, stimulatory at low doses but inhibitory at higher doses (1). In addition, the form, route, and timing of estrogen seem to be important determinants of estrogen effects on growth (2). Pubertal estrogen replacement treatment is customarily delayed until about 15 years of age in the USA to give GH treatment more time to act because standard estrogen treatment inhibits growth (3), in part by direct effects on epiphyseal senescence and fusion (4, 5) and in part by acting as a GH antagonist (6).

Our pilot studies suggest that the form and route of estrogen are important determinants of estrogen effects on growth (2, 7). We recently found that very low doses of parenteral (IM depot) estradiol (E2) together with recombinant growth hormone (GH) to Turner syndrome patients as young as 12-12.9 years of age produced a significantly greater adult height than standard doses of oral conjugated estrogen at this age (7). Thus, very low doses of the natural estrogen (estradiol, E2) administered into the systemic circulation seem optimal for growth stimulation.

Very little data are available about the optimal E2 dose for stimulation of epiphyseal growth and how this may relate to the optimal dosage for accrual of bone mineral density and feminization.

Our recent pilot study started with a depot E2 dose of 0.2 mg; the monthly dose was then increased by 0.2 mg at successive 6-month intervals. The lowest dose (0.2 mg) stimulated height velocity the most. However, it did not stimulate breast development as reliably as the larger doses (≥ 0.4 mg monthly), which were also growth stimulatory although to a lesser extent. We propose to resolve questions about whether these disparities were due to the invariable sequential administration of successively larger doses or the inaccuracy of delivery of such low doses by injection, and also to compare the effects on bone mineral density of the equivalent very low and low doses of E2 delivered by transdermal patch. Transdermal E2 delivery systems are now available for easily and reliably delivering the comparable very low doses of E2 in a form more suitable for routine patient care. The current guidelines recommend starting an E2 starting dose for the induction of puberty (5-12.5 mcg daily) that is about one-tenth to one-eighth of the adult dose (100 mcg daily) (8). However, these guidelines note that it is not established whether various means of patch dose fractionation (e.g., administering a quarter patch overnight or daily or administering whole patches for 7-10 days per month) are equivalent.

Pharmacokinetic study of transdermal E2 in Turner syndrome teens showed absorption of E2 by first order kinetics (9). Steady state was achieved approximately 9 hrs after application of a 37.5 µg patch, and serum concentrations reached a mean of 52.9 ± 17.8 (SD) pg/ml. This demonstrates a rise in plasma estradiol of about 1 pg/ml (3.67 pmol/l) for every 1.0 µg applied to the skin, similar to package insert data in adults. This would suggest that a starting dose of 5-10 ug transdermal E2 daily approximates the 133-266 µg monthly amount of E2 delivered by the 0.2-0.4 mg monthly injections of E2 cypionate.

Our preliminary data support this extrapolation. In n = 3 Turner syndrome patients combining a transdermal E2 dose of 17.8 ± 2.1 (SD) mcg for an average of 14 days a month with GH therapy for 1.0 year showed increases in breast tissue diameter of 1.8 ± 0.3 cm (i.e., breast budding), bone mineral density of 0.067 ± 0.06 gm/cm2 in the lumbar spine, and height velocity of 5.16 ± 1.37 cm/year. The new VLTE2 (14 mcg) patch increases lumbar spine bone mineral density 2.4% at 1 year in post-menopausal women (P <0.001), but no trials have been conducted in children (package insert).

We now propose to move beyond proof of the principle that systemic administration of very low or low dose E2 is efficacious to the practical application of E2 treatment. Our study used IM depot E2 (E2 cyclopentylpropionate, which is two-thirds E2), the very low doses of which required a compounding pharmacy to prepare a stock solution of 1.0 mg/cc. This was helpful with compliance, but not necessarily accurate and certainly not convenient for routine dispensing of prescriptions. Practically, we propose to extrapolate from this experience with parenteral to the readily available and highly acceptable transdermal preparations: the 14 mcg patch worn for 10 days a month delivers an E2 profile approximately equivalent to the 0.2 mg monthly dose of depot E2, and a 25 mcg patch worn for 10 days a month is approximately equivalent to the 0.4 mg monthly dose of depot E2 (7).

ELIGIBILITY:
Inclusion Criteria:

* 60 subjects will be recruited from participating Pediatric Endocrinology Clinics in the United States.
* Subjects will be 11.5-13.0 years of age and must have completed at least 6 months of GH therapy prior to the study.
* Subjects may not have had any estrogen prior to the study. All subjects must be breast stage 1 and euthyroid prior to the study
* Those on thyroid medication will continue the appropriate thyroid replacement therapy during the study.

Exclusion Criteria:

* On estrogen therapy, breast stage 2 or greater, not on GH for at least 6 months.

Ages: 138 Months to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The net change of height velocity between Group 2 and Group 3 and the net change in predicted height between Group 2 and Group 3. | 12 months

SECONDARY OUTCOMES:
Plasma E2 level to document the dose-response effect of the applied prescription and uterine dimensions to quantitate the estrogenic effect on growth and development of the uterus. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rosenfield, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan